CLINICAL TRIAL: NCT07234409
Title: Standard Flank Approach vs Supine Approach for Robot-assisted Partial Nephrectomy
Brief Title: Clinical Trial Addressing the Best Surgical Approach for Partial Nephrectomy With Single Port Robotic System in the Management of Localized Renal Cell Carcinoma
Acronym: K3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 5448_16.04.2025_N_bis
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Kidney Neoplasm
Keywords: kidney cancer; robotic surgery; single port; supine position; full flank position
MeSH Terms: conditions — Kidney Neoplasms; Deception

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A - STANDARD FLANK APPROACH (Other): Patients are positioned laterally (on their side) with the operative flank elevated at a 12-15° angle. The Da Vinci SP robotic system is docked either transperitoneally or retroperitoneally through a single access port.
  Interventions: Other: STANDARD FLANK APPROACH
- GROUP B - Supine anterior retroperitoneal approach (SARA). (Experimental): Patients are positioned supine with a mild Trendelenburg tilt (0°-10°). A retroperitoneal space is created through an anterior incision, providing direct access to the kidney without repositioning.
  Interventions: Procedure: Supine anterior retroperitoneal approach (SARA).

INTERVENTIONS:
Other: STANDARD FLANK APPROACH — Patients are positioned laterally (on their side) with the operative flank elevated at a 12-15° angle. The Da Vinci SP robotic system is docked either transperitoneally or retroperitoneally through a single access port.
  Arms: GROUP A - STANDARD FLANK APPROACH
Procedure: Supine anterior retroperitoneal approach (SARA). — Patients are positioned supine with a mild Trendelenburg tilt (0°-10°). A retroperitoneal space is created through an anterior incision, providing direct access to the kidney without repositioning
  Arms: GROUP B - Supine anterior retroperitoneal approach (SARA).

SUMMARY:
This study aims to find out which surgical position is safer and works better for patients candidate to robot-assisted partial nephrectomy (RAPN) - a minimally invasive procedure to remove a small kidney tumor while preserving healthy kidney tissue.

During this operation, the patient can be placed in two different positions:

* the standard flank position, where the patient lies on their side
* a newer supine position, where the patient lies on their back using a technique called Supine Anterior Retroperitoneal Approach (SARA).

Both approaches are performed using the Da Vinci® Single Port (SP) robotic system, a state-of-the-art surgical robot that allows the operation to be done through a single small incision.

The traditional flank position has been used for many years, but it can be uncomfortable for patients and may increase the risk of certain anesthetic or nerve-related complications, especially in people with higher body weight. The new supine SARA technique could make surgery faster, safer, and less painful, but it has not yet been tested in a randomized study.

This is the first clinical trial designed to directly compare these two approaches in patients with small and localized kidney cancers (tumors ≤7 cm, stage cT1).

The study will include 124 patients treated at ASST Grande Ospedale Metropolitano Niguarda in Milan, Italy - a leading center in robotic urologic surgery.

DETAILED DESCRIPTION:
Study Objectives

Primary Objective:

To compare the outcomes of RAPN performed with the SARA approach versus the standard flank approach in achieving a "trifecta outcome," defined as:

* No intraoperative adverse events;
* Negative (cancer-free) surgical margins;
* Hospital discharge on postoperative day 1.

Secondary Objectives:

* To compare both approaches according to the rate of achievement of two out of three outcomes, and according to each outcome composing the trifecta separately.
* To evaluate postoperative recovery, including pain scores, time to first walk, time to first flatus, total use of pain medication, and readiness for discharge.
* To compare the rates and severity of postoperative complications within 30 days after surgery.
* To assess surgical parameters such as total operative time, ischemia time, and blood loss.
* To analyze functional outcomes, such as kidney function recovery (Δ eGFR at 30 days).

Study Design This is a prospective, single-center, randomized controlled trial conducted at the Department of Urology, ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy.

Eligible participants will be randomly assigned 1:1 to one of two groups:

Group A (Control): Standard flank approach (transperitoneal or retroperitoneal) using the Da Vinci SP system. Patients are positioned laterally (on their side) with the operative flank elevated at a 12-15° angle. The Da Vinci SP robotic system is docked either transperitoneally or retroperitoneally through a single access port. The tumor is resected and kidney reconstruction is performed according to standard RAPN procedures Group B (Experimental): Supine anterior retroperitoneal approach (SARA) using the Da Vinci SP system. Patients are positioned supine with a mild Trendelenburg tilt (0°-10°). A retroperitoneal space is created through an anterior incision, providing direct access to the kidney without repositioning. The same Da Vinci SP system and standard nephron-sparing techniques are used.

Both groups follow identical perioperative protocols for anesthesia, analgesia, and postoperative care.

Population Adults (age 18 or older) with a single kidney tumor measuring up to 7 cm, who are eligible for robotic partial nephrectomy with the Da Vinci SP system, may be invited to participate. Patients with kidney tumor more than 7 cm or advanced tumors infiltrating the surroinding tissues, solitary kidneys, previous kidney surgery on the same kidney, or severe kidney disease will not be eligible.

ELIGIBILITY:
* Age ≥ 18 years;
* Presence of a single, unilateral, primary renal mass ≤ 7 cm in diameter (clinical stage cT1) documented CT scan
* No evidence of systemic disease or lymph node involvement;
* Candidate for robot-assisted partial nephrectomy using the Da Vinci SP platform;
* Signed informed consent
* Absence of solitary kidney status
* No previous partial nephrectomy/ies on the same kidney
* Absence of preoperative chronic kidney disease (CKD) stage 5
* Absence of any condition that makes mandatory or significantly more adequate the choice of a specific approach over the others (e.g., multiple previous major abdominal surgeries, horseshoe kidney, presence of stomas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
TRIFECTA | Intra and perioperative
  Trifecta is defined as the coexistence of these three conditions:
  1. Absence of any intraoperative adverse event
  2. Absence of positive surgical margins
  3. Hospital discharge at postoperative day 1

SECONDARY OUTCOMES:
Partial trifecta achievement | Intra and perioperative
  Secondary end point of the study is to compare RAPN performed with the SARA approach vs RAPN performed with standard flank approach according to the rate of achievement of two out of three outcomes, and lastly according to each outcome composing the trifecta separately.
30 day complications | 30 postoperative days
  complications

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Dell'Oglio, MD PhD, Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda
Locations (1):
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided